CLINICAL TRIAL: NCT06366932
Title: Optimization of Atopic Dermatitis Treatment That Requires Second-line Systemic Therapy Through Multiomic Predictive Models of Treatment Response (DermAtOmics-II)
Brief Title: Optimization of Atopic Dermatitis Treatment That Requires Second-line Systemic Therapy Through Predictive Models
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DermAtOmics-II
Record Dates: First submitted 2024-03-07; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; tralokinumab; upadacitinib; baricitinib; abrocitinib

STUDY DESIGN:
Intervention Model Description: Phase IV, low-intervention clinical trial to develop prediction models that allow to determine the most appropriate therapeutic strategy in patients diagnosed with atopic dermatitis that need second-line systemic treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: patients who are about to initiate treatment (Other): Patients will receive the dose used in routine clinical practice.
  Once the patient is included in the clinical trial their therapeutic management will be conducted according to standard clinical practice, but some additional procedures will be performed:
  1. The frequency of follow-up visits will be increased in order to collect data related to clinical efficacy, safety and quality of life.
  2. Blood samples will be obtained for biochemical, pharmacogenetic and immunological biomarker analysis
  Interventions: Drug: Second-line systemic treatment
- Cohort 2: patients who are already receiving second-line systemic treatment (Other): If the patient is receiving second-line therapy at the moment of the inclusion, data will be collected from clinical records from treatment start until study inclusion and prospectively after study inclusion.
  Interventions: Other: Folllow-up of second-line systemic treatment already started

INTERVENTIONS:
Drug: Second-line systemic treatment — Patients with moderate to severe atopic dermatitis refractory to topical medication, who also have previous experience with cyclosporine and an unsatisfactory response, or in whom the use of cyclosporine is considered inappropriate due to contraindication or intolerance, are candidates for treatment with other alternatives (Dupilumab, Tralokinumab, Upadacitinib, Baricitinib, Abrocitinib).
  Other Names: Dupilumab, Tralokinumab, Upadacitinib, Baricitinib, Abrocitinib
  Arms: Cohort 1: patients who are about to initiate treatment
Other: Folllow-up of second-line systemic treatment already started — If the patient is receiving second-line therapy at the moment of the inclusion, data will be collected from clinical records from treatment start until study inclusion and prospectively after study inclusion.
  Arms: Cohort 2: patients who are already receiving second-line systemic treatment

SUMMARY:
This is a low-intervention phase IV trial. The main objective is to optimize the treatment of patients with moderate-severe atopic dermatitis that require systemic treatment after failure, intolerance or contraindication to cyclosporine.

DETAILED DESCRIPTION:
Primary outcome is the percentage of patients with primary non-response to second-line treatment. Defined as fail to achieve EASI-75 (a 75% improvement in EASI score) at week 16 of follow-up. A 12-month recruitment period is planned and about 150 patients with moderate-severe atopic dermatitis will be recruited. The study is divided into two cohorts. All patients diagnosed with moderate to severe atopic dermatitis who are going to receive second-line systemic treatment at the Dermatology Department of La Paz University Hospital are selected in cohort 1. Patients will receive the starting dose used in routine clinical practice. All patients diagnosed with moderate to severe atopic dermatitis who are receiving second-line systemic treatment at the Dermatology Department of La Paz University Hospital will be selected in cohort 2.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

1. Subjects diagnosed with moderate-severe atopic dermatitis who are going to receive an authorized second-line systemic treatment.
2. Participants must be willing and able to provide written informed consent prior the initiation of any study procedures.
3. For children, parent/legal guardian must provide written informed consent. If age >11 years old, the minor must give assent.
4. Participant is willing and able to adhere to the procedures specified in this protocol.

Cohort 2:

1. Subjects diagnosed with moderate-severe atopic dermatitis who are already receiving authorized second-line systemic therapy at the time of selection.
2. Participants must be willing and able to provide written informed consent prior the initiation of any study procedures.
3. For children, parent/legal guardian must provide written informed consent. If age >11 years old, the minor must give assent.
4. Participant is willing and able to adhere to the procedures specified in this protocol.

Exclusion Criteria:

1. Any investigational drug within 60 days prior to study drug administration.
2. Any condition or situation precluding or interfering the compliance with the protocol.
3. Women of childbearing potential must have a negative urine pregnancy test at Screening and Day 0.
4. Women of childbearing potential must commit not to become pregnant. They must be willing to use highly effective contraceptive methods or have practiced sexual abstinence during the study. Highly effective contraceptive methods include oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation; intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; vasectomised partner and sexual abstinence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with primary non-response to second-line treatment. | Week 16
  Fail to achieve EASI-75 (a 75% improvement in Eczema Area and Severity Index [EASI] score). The minimum EASI score is 0 and the maximum EASI score is 72.

SECONDARY OUTCOMES:
Percentage of patients achieving EASI-75 | Week 6
  Fail to achieve EASI-75 (a 75% improvement in Eczema Area and Severity Index [EASI] score). The minimum EASI score is 0 and the maximum EASI score is 72.
Time to treatment failure after week 16 | Week 16
  Time to treatment failure with cyclosporine defined as Eczema Area and Severity Index (EASI) ≤ 50 during follow-up after week 16.
Mean percentage of change in Eczema Area and Severity Index (EASI) score | Week 16
  Mean percentage of change in EASI score from baseline to week 16.
Percentage of change in SCORAD (SCORing Atopic Dermatitis) | Week 16
  Is the score of the severity of atopic dermatitis. It includes the evaluation of the affected areas. The intensity of the lesions and the subjective symptoms of the patient. Classifies AD as Mild >25, Moderate 25-50, and Severe >50
Improvement of at least 75% in SCORAD (SCORing Atopic Dermatitis) | Through study completion, an average of 1 year
  Percentage of patients experiencing an improvement of at least 75% in SCORAD from the baseline value.
  The SCORAD for that individual is A/5 + 7B/2 + C. The total area is 'A', which has a possible maximum of 100%. The intensity scores are added together to give 'B' (maximum 18). The subjective symptoms is 'C' (maximum 20).
Change of IGA (Investigator Global Assessment) | Week 16
  Investigator Global Assessment (IGA) is a simple objective measure providing an overall evaluation. It uses a 5-point scale (clear=0; almost clear=1; mild=2; moderate=3; severe=4).
Time to IGA score of 0/1 (Investigator Global Assessment) | Through study completion, an average of 1 year
  Time to IGA score of 0/1 (clear or almost clear).
Change of BSA (Body surface area) | Week 16
  Change of BSA (Body surface area) involment
Change in NRS | Week 16
  Change in NRS (numerical rating scale). The NRS is comprised of one item and represents the numbers 0 ("no itch") to 10 ("worst imaginable itch").
Change in RECAP | Week 16
  RECAP (Recap of atopic eczema) is used to assess the control of different degrees of eczema severity through 7 items.
Percentage of patients having a variation of 4 points in their improvement in DLQI | Through study completion, an average of 1 year
  Dermatology Life Quality Index is a validated and widely used 10-item questionnaire with paediatric versions (0-3 and 4-16 years). A variation of 4 points is considered a clinically meaningful endpoint.
Change in POEM (Patient-Oriented Eczema Measure) | Week 16
  The Patient-Oriented Eczema Measure (POEM): is a validated tool in which the patient self-assesses how many days they experienced seven distinct items (itch, sleep disturbance, bleeding, weeping/oozing, cracking, flaking, dryness of the skin) during a period of 1 week. The maximum score is 28 points.
Rate of adverse events associated to second-line systemic treatment | Through study completion, an average of 1 year
  Any untoward medical occurrence in a patient or clinical trial participant, which does not necessarily have a causal relationship with the research procedures or the investigational medicinal product.
Percentage of patients reaching EASI-90 (Percentage of patients reaching 90 percentage) | Through study completion, an average of 1 year
  Percentage of patients reaching 90 percentage (EASI-90) improvement from baseline during follow-up. The minimum EASI (Eczema Area and Severity Index) score is 0 and the maximum EASI score is 72.

CONTACTS AND LOCATIONS:
Overall Officials: Irene García, MD, Principal Investigator — Hospital La Paz
Locations (1):
- Hospital La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No